CLINICAL TRIAL: NCT03281239
Title: Study of the Impact of Welding Fumes on the Arterial System : RISCAS Study
Acronym: RISCAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the difficulties of inclusion, it was decided not to extend this period
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC17.0131 RISCAS
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Effects of Welding Fumes Components
Keywords: welder, airport agent, Welding fumes
MeSH Terms: interventions — Hematologic Tests; Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- welder/airport agent (Experimental): No drug and no placebo were used in this study.
  Interventions: Diagnostic Test: Laser doppler, blood tests, and holter ECG

INTERVENTIONS:
Diagnostic Test: Laser doppler, blood tests, and holter ECG — Diagnostic tests :
  * laser doppler
  * blood tests
  * Holter ECG. No drug and no placebo were used in this arm.

SUMMARY:
Metals and oxydes are found in welding fumes and are thought to participate in increasing cardiovascular risk in exposed workers. Investigators aimed to evaluate the impact of this occupational exposure on cardiovascular system in a highly exposed population, ship repairing welders and to compare this population to paired controls.

DETAILED DESCRIPTION:
In an exposed-non-exposed study, investigators will include 30 welders and 30 airport runway agents for control. As part of cardiovascular independent risk factors, microvascular endothelial function will be evaluated directly by laser Doppler flowmetry. Blood samples will be also collected and circulating markers of endothelial function (VW factor, E-selectin, VCAM, ICAM, circulating DNA), inflammation (CRP, IL-1β, IL-8, TNFα, IL-10), platelet activation (procoagulant microparticles, thrombin generation, fibin monomer) will be measured. A complete clinical and functional cardiovascular status will be documented in every participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years
* Employee performing welding or airport operations
* free, informed and written consent
* Being affiliated to a social security system

Exclusion Criteria:

* Taking cardiovascular medications which modify endothelial function and / or coagulation (antiplatelet, antihypertensive, cardiotropic).
* People with a history of ischemic cardiovascular disease, thrombotic disease, chronic inflammatory disease
* Pregnant women
* People with health status would be likely, in the baseline state, to have parameters studied in the study disrupted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Vascular reactivity | 1 day
  Assessement of microvascular reactivity by laser Doppler flowmetry associated to iontophoretic administration of ACh and SNP

SECONDARY OUTCOMES:
Coagulation activation | 1 day
  Assessment of markers of blood coagulation
vascular inflammation | 1 day
  Assessment of factors of inflammation
Impregnation of metals activation | 1 day
  Assessment of impregnation factor
Oxidative stress activation | 1 day
  Assessment of markers of oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France